CLINICAL TRIAL: NCT01887613
Title: Specified Drug Use-Results Survey of Regnite
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: REG001
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Restless Legs Syndrome
Keywords: Gabapentin
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Regnite group: Patients who receive Regnite
  Interventions: Drug: Regnite

INTERVENTIONS:
Drug: Regnite — oral
  Other Names: gabapentin enacarbil

SUMMARY:
This study is to investigate the long-term safety and efficacy and the information on the proper use of Regnite® under conditions of daily clinical use.

DETAILED DESCRIPTION:
Sleeping condition and severity of restless legs syndrome (RLS) were recorded at the start and during the treatment. The treatment period is scheduled to last 52 weeks in principle. For patients completing or discontinuing the use of Regnite® within 52 weeks, follow up on the withdrawal and rebound syndrome will be conducted up to 4 weeks of completion or discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe idiopathic restless legs syndrome

Exclusion Criteria:

* Patients with a history of hypersensitivity to any ingredients in Regnite or gabapentin
* Patients with severely impaired renal function (creatinine clearance of less than 30 mL/min)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate to severe idiopathic restless legs syndrome
Sampling Method: Non-Probability Sample
Enrollment: 1597 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Safety such as occurrence of adverse drug reactions and lab-tests | Up to 52 weeks

SECONDARY OUTCOMES:
Restless Leg Syndrome score | Baseline and at 52 weeks
Clinical Global Impression | Baseline and at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku